CLINICAL TRIAL: NCT03500042
Title: Effects of Different Modes of Respiratory Muscular Threshold Loads Training on Respiratory Mechanics and Neural Respiratory Drive(NRD) in Patient With Stable Chronic Obstructive Pulmonary Disease(COPD).
Brief Title: Effects of Different Modes of Respiratory MuscleTraining on Respiratory Mechanics and NRD in Patient With Stable COPD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-HXNK-008
Record Dates: First submitted 2018-03-26; First posted 2018-04-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; inspiratory muscle training; expiratory muscle training; Neural Respiratory Drive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- respiratory muscle weakness (Experimental): Patients with respiratory muscle weakness are performing the inspiratory pressure threshold device, expiratory pressure threshold device and concurrent inspiratory and expiratory muscle device for one minute randomly.
  Interventions: Device: inspiratory pressure threshold device
- normal respiratory muscle (Experimental): Patients with respiratory muscle weakness are performing the inspiratory pressure threshold device, expiratory pressure threshold device and concurrent inspiratory and expiratory muscle device for one minute randomly.
  Interventions: Device: inspiratory pressure threshold device

INTERVENTIONS:
Device: inspiratory pressure threshold device — The threshold loading device is composed of a mouth -piece attached to a small plastic cylinder that contains a spring-loaded poppet value. The valve opens to permit inspiratory flow only once the person has generated adequate negative intrathoracic pressure to condense the spring.
  Other Names: expiratory pressure threshold device; concurrent inspiratory and expiratory muscle device

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic respiratory disease characterized by persistent airflow limitation. The patients are suffering dyspnea year by year, resulting in the decreased exercise tolerance and quality of life. Patients with COPD often have both inspiratory muscles and expiratory muscle dysfunction. Respiratory muscle training was one of the widely used pulmonary rehabilitation method in COPD patients. Respiratory muscle training include inspiratory training ,expiratory training and concurrent inspiratory and expiratory muscle training . Both of the training methods are effective. However, the effects of these different types of respiratory muscle training method on the respiratory physiology and neural respiratory drive of COPD are still unclear. Therefore, the purpose of this study was to investigate the different effects of these respiratory muscle training methods on respiratory mechanics and central drive in COPD patients. Besides,the effect of the different respiratory muscle training methods was compared between patients with and without respiratory muscle weakness.

DETAILED DESCRIPTION:
The patients with COPD will participate in a rehabilitation program including inspiratory muscle training, expiratory muscle training and concurrent inspiratory and expiratory muscle training.

The outcome measures are the classic respiratory mechanics indicators and respiratory center drive.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary function test of forced expiratory volume at one second (FEV1)/forced vital capacity(FVC) < 70% after inhalation of bronchial dilation agent. Patients in a clinically stable state.

Exclusion Criteria:

* Patients were excluded if they had other respiratory diseases ,or evidence of pneumothorax or mediastinal emphysema and pacemaker installed.

Patients with acute cardiovascular event and severe cor pulmonale. Patients with poor compliance. An Other causes of diaphragmatic dysfunction

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic function | Change from baseline in diaphragm electromyogram at the load of threshold (10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  Diaphragmatic function can be assessed by diaphragm electromyogram(EMGdi) which reflect the physiological activity of the diaphragm and indicate functional status of the central drive.

SECONDARY OUTCOMES:
Respiratory pressure | Change from baseline in respiratory pressure at the load of threshold (10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  Respiratory pressure parameter is transdiaphragmatic pressure ( Pdi) in cmH2O, which reflect the strength of diaphragm.
Respiratory volume | Change from baseline in respiratory volume at the load of threshold (10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  Respiratory volume parameter is minute ventilation (VE) in liter(L).
respiratory work | Change from baseline in transdiaphragmatic pressure time product at the load of threshold (10 minutes later,20minutes later,30 minutes later, 40 minutes later)
  respiratory work is associated with transdiaphragmatic pressure time product

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No